CLINICAL TRIAL: NCT00889707
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study of Transperineal Intraprostatic Injection of PRX302 for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Transperineal Intraprostatic Injection of PRX302 Under Ultrasound Guidance for Management of Prostatic Hyperplasia
Acronym: TRIUMPH-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRX302-2-03
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; BPH; Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — PRX302

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Drug (Experimental): PRX302
  Interventions: Drug: PRX302
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRX302 — PRX302 will be administered at a volume equivalent to 20% of the prostate volume and at a fixed concentration. Treatment will be administered through 1 injection into the transition zone of each lobe of the prostate. A minimum of 2 deposits will be made in the transition zone into each of the right and left lobes of the prostate, with a minimum of 1.0 mL per deposit.
  Arms: Active Drug
Drug: Placebo — PRX302 will be administered at a volume equivalent to 20% of the prostate volume and at a fixed concentration. Treatment will be administered through 1 injection into the transition zone of each lobe of the prostate. A minimum of 2 deposits will be made in the transition zone into each of the right and left lobes of the prostate, with a minimum of 1.0 mL per deposit.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PRX302 is safe and effective in the treatment of moderate to severe Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study of transperineal intraprostatic injection of PRX302 under sonographic guidance. Subjects will be randomly assigned to the two treatment groups in a ratio of 2:1 between PRX302 and Placebo, stratified by prostate size and baseline IPSS.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 40 to 80 years;
* Lower urinary tract symptoms (LUTS), such as frequency, nocturia, urgency, weak urine stream, hesitancy, intermittency or post-void dribbling attributable to BPH for at least 6 months prior to dosing;
* Untreated, intolerant or refractory to α-blockers; should not have received the medication for at least 2 weeks prior to screening and 4 weeks prior to dosing;
* Subjects with PSA values 4 - 10 ng/mL should be assessed or medical records checked (e.g. biopsy report) to rule out the presence of prostate cancer;
* Untreated, intolerant or intolerant to 5-α reductase inhibitors AND must be off medication for at least 6 months prior to dosing;
* IPSS of 15 or higher;
* Prostate volume at screening estimated at 30 to 100 mL as determined by TRUS;
* Provided written Informed Consent for participation in the study.

Exclusion Criteria:

* Maximum urine flow rate (Qmax) of greater than 12 mL/sec;
* Inability to void at least 150 mL of urine;
* Post voiding residual urine volume (PVR) of greater than 200 mL;
* Subjects unable to stand to void;
* Subjects with acute or chronic bacterial prostatitis;
* Using drugs (e.g. estrogen, androgen) that can produce androgen depression or anabolic steroids;
* Penile prosthesis or artificial urinary sphincter;
* Presence of prostatic cyst larger than 1 cm in diameter;
* Unwilling to use condoms for 3 weeks post-treatment to prevent pregnancy and to avoid semen contact with partner(s);
* Urethral stricture disease;
* Bladder neck abnormalities/strictures;
* Significant median lobe hyperplasia that contributes to outflow obstruction;
* Confirmed or suspected neurogenic bladder dysfunction;
* Systemic neurological disorders that may affect voiding function;
* Previous pelvic surgery, trauma or radiation;
* Active genitourinary infection within 7 days before screening;
* Significant renal dysfunction (as evidenced by a serum creatinine > 1.6 mg/dL on the screening laboratory evaluation);
* Abnormal liver function as evidenced by any of the following abnormal laboratory values being greater than 1.5 upper limit of normal (ULN) at screening:

  * alkaline phosphatase (ALP);
  * total bilirubin;
  * alanine transferase (ALT); and/or
  * aspartate aminotransferase (AST);
* Abnormal Prothrombin Time (PT > 13 sec) / International Normalized Ratio (INR > 1.2);
* Severe cardiovascular or hepatic disease (American Society of Anesthesiologists [ASA] > 3); Presence of suspected or confirmed malignancy other than non-melanomatous, cutaneous malignancies which have undergone curative interventions;
* Receiving anticoagulants (Subjects receiving anticoagulants may be enrolled after discontinuation of anticoagulant therapy and return of INR level to within normal limits (INR < 1.2) before dosing day. Subjects receiving platelet inhibitors (including garlic) must be off the inhibitors for at least 6 days or more. Subjects unable to discontinue anticoagulant therapy may not be enrolled in this study);
* Subjects who have received any treatment for BPH other than α-blockers, 5-α reductase inhibitors or phytotherapy;
* Subjects taking α-blockers and phytotherapy within 2 weeks of screening and 4 weeks of dosing;
* Subjects receiving 5-α reductase inhibitors within 6 months of dosing;
* Subjects taking part in other experimental programs prior to the start of the study or during the study period;
* Any medical, psychological or other condition or medical history of the subject that, in the opinion of the Investigator or the Sponsor's Medical Monitor, unduly increases the risk of subject's participation or that would unnecessarily confound the data to be collected in this study;
* Unable or unwilling to comply with the requirements of the protocol.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pommerville, MD, Principal Investigator — CanMed Clinical Reaearch Inc.; Mostafa Elhilali, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (9):
- Canada (9):
  - Andreou Research, Surrey, British Columbia
  - CanMed Clinical Research Inc., Victoria, British Columbia
  - Dr. Steinhoff Clinical Research, Victoria, British Columbia
  - Bramalea Medical Centre, Brampton, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Urology Associates / Urology Medical Research, Kitchener, Ontario
  - The Fe/Male Health Centers, Oakville, Ontario
  - Anthony Skehan Medicine Professional Corp., Thunder Bay, Ontario
  - McGill University Health Centre, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Targeted patient enrollment was 90. 92 patients were actually randomized and dosed before enrollment was discontinued.
Groups:
- PRX302: 0.6 microgram/gram prostate weight in 2% (weight/volume) human serum albumin (HSA)
- Placebo: 2% (weight/volume) human serum albumin (HSA) without PRX302
Period: Overall Study
Arm/Group | PRX302 | Placebo
Started | 61 | 31
Completed | 54 | 21
Not Completed | 7 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 2 | 5

BASELINE CHARACTERISTICS:
Population: All randomized patients who received study drug.
Groups:
- PRX302: 0.6 microgram/gram prostate in 2% HSA
- Placebo: 2% HSA without PRX302
- Total: Total of all reporting groups
Arm/Group | PRX302 | Placebo | Total
Number analyzed (Participants) | 61 | 31 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 17 | 52
  >=65 years | 26 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.74) | 63.5 (8.36) | 63.6 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 31 | 92
Region of Enrollment [Number; unit: participants]
  Canada | 61 | 31 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in International Prostate Symptom Scale (IPSS) of Lower Urinary Tract Symptoms From Baseline to 3 Months (Total Score at 3 Months Minus Total Score at Baseline)
Description: Total of 7 questions regarding lower urinary tract symptoms, with each question scored on a range of 0 (not at all) to 5 (almost always have the symptom). The total score is the summation of all 7 questions, and therefore has a possible range of 0 to 35.
Time Frame: 3 months post-treatment
Population: The efficacy evaluable (EE) protocol defined primary analysis population, defined as (1) all patients who received the randomized treatment in full, (2) completed the Month 3 efficacy assessments, and (4) did not have a major protocol deviation that could confound the assessment of efficacy as determined by a blinded, independent data review panel.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | PRX302 | Placebo
Number analyzed (Participants) | 52 | 21
score | -9.1 (5.95) | -5.8 (5.40)
Statistical Analysis 1: Comparison: PRX302 vs Placebo; Test type: Superiority or Other; p = 0.040, ANCOVA — Test of superiority computed using an ANCOVA model with terms for treatment group, baseline total IPSS, and baseline prostate volume. Tested for 2-sided 0.05 level of statistical significance; ANCOVA model with terms for treatment group, baseline total IPSS, and baseline prostate volume

2. Secondary Outcome: Change in Maximum Urinary Flow Rate (Qmax) From Baseline to 3 Months (Qmax at 3 Months Minus Qmax at Baseline)
Description: A printout of uroflowmetry was provided to a central, blinded, independent reviewer for determination of the Qmax values to be used for evaluation of efficacy. The central, independent, blinded reviewer determined the Qmax from over-reads of the uroflowmetry printouts, applying the 2-second rule to reduce variability and increase the accuracy.
Time Frame: 3 months after treatment
Population: The protocol-defined efficacy evaluable (EE) primary analysis population, defined as (1) all patients who received the randomized treatment in full, (2) completed the Month 3 efficacy assessments, and (4) did not have a major protocol deviation that could confound the assessment of efficacy as determined by a blinded, independent data review panel
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | PRX302 | Placebo
Number analyzed (Participants) | 52 | 21
ml/sec | 3.13 (4.35) | 1.31 (3.16)
Statistical Analysis 1: Comparison: PRX302 vs Placebo; Test type: Superiority or Other; p = 0.047, ANCOVA — ANCOVA model with terms for treatment group, baseline total IPSS, baseline prostate volume, and baseline Qmax; Model with terms for treatment group, baseline total IPSS, baseline prostate volume, and baseline Qmax

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PRX302 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/31
Other Adverse Events (participants affected / at risk) | 38/61 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX302 (N=61) | Placebo (N=31)
Medical Device Pain (General disorders) | 1 (1) | 0 (0)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX302 (N=61) | Placebo (N=31)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Dysuria (Renal and urinary disorders) | 18 (18) | 2 (2)
Haematuria (Renal and urinary disorders) | 18 (18) | 11 (11)
Micturition Urgency (Renal and urinary disorders) | 14 (14) | 3 (3)
Nocturia (Renal and urinary disorders) | 2 (2) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 15 (15) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Haematospermia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Perineal Pain (Reproductive system and breast disorders) | 9 (9) | 0 (0)
Prostatic Pain (Reproductive system and breast disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators will take all steps reasonably necessary to hold Protox's Proprietary Information in trust and confidence, will not use Proprietary Information in any manner or for any purpose not expressly set forth in their Agreement, and will not disclose any such Proprietary Information to any third party without first obtaining Protox's express written consent.